CLINICAL TRIAL: NCT06515405
Title: Effect of Early Hydrocortisone on Risk of Gastrointestinal Perforations in Extremely Preterm Infants: A Protocol for a Retrospective Cohort Study Using Routinely Collected Data
Brief Title: Effect of Early Hydrocortisone on Risk of Gastrointestinal Perforations in Extremely Preterm Infants
Status: Active, not recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 293603
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Intestinal Perforation
Keywords: Preterm Infant; Hydrocortisone
MeSH Terms: conditions — Intestinal Perforation; Premature Birth | interventions — Hydrocortisone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Not exposed to early hydrocortisone
  Interventions: Drug: Hydrocortisone
- Exposed to early hydrocortisone
  Interventions: Drug: Hydrocortisone

INTERVENTIONS:
Drug: Hydrocortisone — Cohort members will be considered to be exposed to early hydrocortisone if either:
  1. They receive early hydrocortisone started on postnatal day 1 or 2 and given for more than seven consecutive days OR
  2. They receive early hydrocortisone started on postnatal day 1 or 2 and are being cared for in a PROHYDRO unit but die on or before postnatal day 8.
  PROHYDRO units are defined as units who, at the time the baby was born, had implemented a protocol for use of prophylactic hydrocortisone as part of routine care for babies born less than 28 weeks' gestation. A unit may change from being a non-PROHYDRO unit to a PROHYDRO unit if a new early hydrocortisone protocol is introduced during the study period (2016-2023).

SUMMARY:
A large, randomised control trial, the PREMILOC trial, has established that giving low dose hydrocortisone prophylactically in the first ten days of life reduces the risk of bronchopulmonary dysplasia in babies born before 32 weeks' gestation. However, the PREMILOC trial was underpowered to investigate rarer side effects, such as gastrointestinal perforation. This study aims to establish whether the odds of gastrointestinal perforation increase when extremely preterm infants are given prophylactic hydrocortisone in the first ten days of life.

This retrospective cohort study will use routinely collected data from the U.K. National Neonatal Research Database. The investigators will examine the records of all infants born before 28 weeks' gestation and cared for in English and Welsh neonatal units between 2016 and 2023. Infants will be considered exposed if they received hydrocortisone for at least eight consecutive days, beginning on postnatal day 1 or 2. The primary outcome will be gastrointestinal perforation, as recorded in the infant's neonatal unit record. This outcome will be validated with the original care teams for a sample of babies. Data will be analysed using a propensity score matched approach to reduce the impact of confounding.

ELIGIBILITY:
Inclusion Criteria:

Infants who:

* were admitted to a neonatal unit between the 1st January 2016 and 31st March 2023 and
* received any of their care in a NHS neonatal unit in England and Wales (part of UK Neonatal Collaborative and therefore contributing data to the NNRD) and
* were born before 28 weeks' gestation.

Exclusion Criteria:

* They have missing data for principal background variables (gestational age at birth, birth weight, year of birth and date of death for those that died).
* Their recorded birthweight absolute value z score exceeds 4 or is missing.
* They died on postnatal day 1 or 2 .

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Infants born before 28 weeks' gestation and admitted to English and Welsh neonatal units.
Sampling Method: Non-Probability Sample
Enrollment: 16000 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal (GI) perforation | From date of birth until day 14 of life
  A baby will be considered to have had a gastrointestinal perforation if their National Neonatal Research Database record includes a record of a GI perforation in the diagnoses field.

SECONDARY OUTCOMES:
Survival without gastrointestinal perforation | From date of birth until the date of discharge from final neonatal unit, assessed up to 24 months
  Baby survived to discharge from neonatal unit without a gastrointestinal perforation
Mortality before discharge home | From date of birth until the date of discharge from final neonatal unit, assessed up to 24 months
  Baby died before discharge from neonatal unit
Total length of stay | From date of birth until the date of discharge from final neonatal unit, assessed up to 24 months
  Length of stay in neonatal care
Proportion of days on unit being mechanically ventilated | From date of birth until the date of discharge from final neonatal unit, assessed up to 24 months
Bronchopulmonary dysplasia | From date of birth until 36 weeks' postmenstrual age (PMA)
  any respiratory or ventilatory support or supplemental oxygen at 36 weeks' postmenstrual age (PMA)
Bronchopulmonary dysplasia | From date of birth until 36 weeks' postmenstrual age (PMA)
  Using an adapted Jensen criteria based on the highest level of respiratory support at 36 weeks PMA

OTHER OUTCOMES:
Necrotising enterocolitis | From date of birth until the date of discharge from final neonatal unit, assessed up to 24 months
  UK National Neonatal Audit Programme definition
Severe necrotising enterocolitis | From date of birth until the date of discharge from final neonatal unit, assessed up to 24 months
  Necrotising enterocolitis confirmed at surgery or post-mortem or stated as cause of death
Pragmatically defined necrotising enterocolitis | From date of birth until the date of discharge from final neonatal unit, assessed up to 24 months
  a recorded diagnosis of necrotising enterocolitis and received at least 5 consecutive days of antibiotics whilst also nil by mouth
Late onset sepsis | From postnatal day 3 until the date of discharge from final neonatal unit, assessed up to 24 months
  One or more episodes of a positive blood or cerebrospinal fluid culture with either a pure or mixed growth of a known pathogenic organism after the first three days following birth
Brain injury occurring at or soon after birth | From date of birth until the date of discharge from final neonatal unit, assessed up to 24 months
  Intracranial haemorrhage, perinatal stroke, central nervous system infection, kernicterus (bilirubin encephalopathy), periventricular leukomalacia or any recorded seizure
Treated retinopathy of prematurity | From date of birth until the date of discharge from final neonatal unit, assessed up to 24 months
  Cryotherapy, laser therapy or injection of anti-vascular endothelial growth factor therapy for ROP in either or both eyes

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Study protocol available now. Analysis code will be available after publication of results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-17): https://cdn.clinicaltrials.gov/large-docs/05/NCT06515405/Prot_SAP_000.pdf